CLINICAL TRIAL: NCT06271226
Title: The Effect of Acupressure Applied to Intensive Care Patients on Pain and Physiological Parameters
Brief Title: The Effect of Acupressure Applied to Icu on Pain and Physiological Parameters
Acronym: EFFECTOFACU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Emine Yaman Lezki, expert nurse, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: OMUKAEK 2022/75; OMUKAEK 2022/75 (Other: ONDOKUZ MAYIS UNIVERSTY)
Record Dates: First submitted 2023-09-19; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Intensive Care Patients; Pain
Keywords: acupressure; critical care nursing; complementary therapies; pain management
MeSH Terms: conditions — Pain; Agnosia | interventions — Acupressure; Control Groups

STUDY DESIGN:
Intervention Model Description: Since there will be variability in patient admissions to intensive care units, block randomization will be used. Three different groups will be coded with different letters (A,B,C) and blocks will be created. Then randomization will be performed by assigning random numbers on the computer. The letters determined in the randomization will be written in closed envelopes and stored, and the randomization process will be carried out by an independent researcher. After the patient who meets the inclusion criteria is identified, the independent researcher will be contacted to find out which group the patient is in.
Who Masked: Participant, Outcomes Assessor
Masking Description: participant and statistical analysis expert is blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- acupressure (Experimental): Information about the pre-procedure intervention will be given. Before acupressure, the participant's physiological parameters and pain score will be recorded, then the hands will be washed in preparation for the acupuncture application and the patient will be placed in a supine or semi-sitting position. Compression points are HT7, P6, P7, Li4, Lv3 points and the location will be determined by the patient's own finger size. Before pressing, a relaxing-relaxing patting motion will be applied to these points for 10 seconds. Then, 1.5 minutes, 5 seconds of thumb pressure and 1 second of free pressure to each point will be applied to each point twice a day (morning and evening). In total it will take 15 minutes to press all the dots. At the end of the application and 15 minutes and 30 minutes after the application, the participant's physiological parameter data and pain score will be re-evaluated and recorded. These data will be recorded twice a day (morning and evening) for 2 days.
  Interventions: Other: acupressure
- plasebo acupressure (Active Comparator): In the placebo group, the preparations and forms applied to the experimental group will be applied in the same way, but in accordance with the literature, an area 1.5 cm away from the acupressure point that has no connection with the acupressure point will be selected and the application will be made in the form of light touch.
  Interventions: Other: placebo acupressure
- control group (Other): During the study, pain and physiological parameters will be monitored and recorded twice a day (morning and evening) for 2 days, without any application (other than the routine treatment given by the physician).
  Interventions: Other: control group

INTERVENTIONS:
Other: acupressure — With acupressure, massage or pressure is applied to certain points on the body with fingers, hands or palms. The pressed points are the points on the skin that are sensitive to bioelectrical impulses and can easily transmit them.
  Other Names: finger pressure
  Arms: acupressure
Other: placebo acupressure — n the placebo group, the preparations and forms applied to the experimental group will be applied in the same way, but in accordance with the literature, an area 1.5 cm away from the acupressure point that has no connection with the acupressure point will be selected and the application will be made in the form of light touch
  Other Names: sham acupressure
  Arms: plasebo acupressure
Other: control group — During the study, pain and physiological parameters will be monitored and recorded twice a day (morning and evening) for 2 days, without any application (other than the routine treatment given by the physician).
  Other Names: follow up
  Arms: control group

SUMMARY:
The aim of this experimental study is to determine the effect of acupressure applied to intensive care patients on pain and physiological parameters (blood pressure, heart rate, respiration and oxygen saturation).

The main questions that the study aims to answer are:

Acupressure applied to intensive care patients has no effect on pain. Acupressure applied to intensive care patients has an effect on pain. Acupressure applied to intensive care patients has no effect on physiological parameters.

Acupressure applied to intensive care patients has an effect on physiological parameters.

Participants will be included in the study after obtaining consent from patients who were treated in the intensive care unit, who scored 9 and above on the glaskow coma scale by evaluating their consciousness status, and had pain after evaluating their pain.

DETAILED DESCRIPTION:
This study is planned to be conducted as a single-blind randomized placebo-controlled-experimental. Patients for randomization will be divided into three groups as experimental, control and plesobo (without true acupressure).

Before the patients in the intensive care unit are included in the study, the state of consciousness with the Glasgow coma scale (GCS) and their pain will be evaluated with the pain scale. Patients with a GCS of 9 and above and who have pain will be included in the study.

Acu points to be used in the study: HT7, P6, P7, Li4, Lv3 points. Li4 and Lv3 are often associated with pain; HT7, P6 and P7 points are especially related to the heart and pericardium.

In the first session of the acupressure intervention to be applied to the experimental group, the patients will be informed about how to perform the application. In order to ensure the physical comfort of the patient, the intervention times will be determined with two application intervals of 4 hours. Physiological parameters and pain score of the experimental group will be recorded before the procedure, then hands will be washed in line with the preparation for acupressure application, and supine or semifowler position will be given according to the patient's preference, taking into account the privacy of the patient. Pressure points will be determined using the patient's own finger measurements.

Before pressing, a relaxing-relaxing patting motion will be applied to these points for 10 seconds. Afterwards, pressure will be applied to each point twice a day (morning and evening) with the thumb for 1.5 minutes, with 5 seconds of pressure and 1 second of free pressure on each point. It will take 15 minutes to press all points in total. At the end of the application and at 15 minutes and 30 minutes after the application, the participant's physiological parameter data and pain score will be re-evaluated and recorded. These data will be recorded 2 times a day (morning and evening) for 2 days.

In the placebo group, the preparations and forms applied to the experimental group will be applied in the same way, but in accordance with the literature, an area 1.5 cm away from the acupressure point that has no connection with the acupressure point will be selected and the application will be made in the form of light touch.

In the control group, pain and physiological parameters will be monitored and recorded twice a day (morning and evening) for 2 days without any application during the study (except for the routine treatment given by the physician).

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years or older
* Volunteering to participate in the research.
* Getting a score of 9 and above on the Glasgow Coma Scale and being able to communicate meaningfully,
* Oxygen saturation of 85 and above
* Mean arterial pressure of 65 mmHg and above

Exclusion Criteria:

* Diagnosis of suspected acute stroke bleeding
* Taking antihypertensive and beta-blocker drugs the start of the study
* Receiving sedation (dormicum, propofol, brunette)
* Presence of ulcers, bilateral paralysis, necrotic tissue and signs of infection (fever, redness, discharge, temperature) at the pressure points
* Situations that will cause the participant to leave the study (death, transfer to another unit, discharge or unwillingness to continue working)
* Receiving inotropic therapy (dopamine, steradine, etc.)
* Absence of analgesic therapy in routine treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
neurological evaluation | it is applied to the participants before the start of the study
  It will be evaluated using the Glaskow Coma scale. With the Glaskow Coma scale, three main functions of the patients, namely eye opening, verbal and motor, are evaluated and scored. Patients' eye opening is scored as 1-4 points, verbal response as 1-5 points, and motor response as 1-6, and the level of consciousness is determined by the total score. As the score of the scale increases, the risk of mortality decreases and the level of awareness increases.
evaluation of pain | The pain scores of the patients included in the study will be recorded twice a day (morning and evening).
  Visual Analog Scale is a one-dimensional measurement tool used to evaluate the pain perceived by the person. The scale is 0-10 cm or 0-100 mm, with no pain (0) at one end, and the worst possible pain (10) at the other end.In the evaluation of VAS, 0 cm = no pain, 0.5-3 cm = mild pain, 3.5-6.5 cm = moderate pain, 7-10 cm = severe pain.
evaluation of physiological parameters | The data of the patients included in the study will be recorded twice a day (morning and evening).
  the physiological parameter was recorded with the registration form.This form includes the patients' blood pressure, heart rate, respiration and SPO2 values.

SECONDARY OUTCOMES:
evaluation of physiological parameters | The data of the patients included in the study will be recorded twice a day (morning and evening) for 2 days.
  blood pressure,heart rate,number of breaths,oxygen saturation

CONTACTS AND LOCATIONS:
Overall Officials: emine yaman lezki, Principal Investigator — Ondokuz Mayıs universty
Locations (1):
- Giresun Eğitim Araştırma Hastanesi, Giresun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
study results can be shared at the end of the study
Supporting Information: Study Protocol, CSR
Time Frame: study results can be shared at the end of the study
Access Criteria: when the study is concluded, the data can be accessed within the limits determined by the principal investigator.